CLINICAL TRIAL: NCT07077499
Title: Analysis of the Cleaning Effect of Pulsed Vacuum Cleaning and Disinfection Device on Rigid Endoscopic Instruments
Brief Title: Cleaning Efficacy of Pulsed Vacuum Device on Rigid Endoscopic Instruments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xue Wang (Other)
Responsible Party: Sponsor-Investigator, Xue Wang, Principal investigator, Shijiazhuang Obstetrics and Gynecology Hospital
Organization: Shijiazhuang Obstetrics and Gynecology Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024039
Record Dates: First submitted 2025-07-05; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Post-Surgical Contamination of Rigid Endoscopic Instruments

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed Vacuum Cleaning Group (Experimental): A total of 400 rigid endoscopic instruments were cleaned using a pulsed vacuum cleaning and disinfection device following manual pre-treatment. The process integrated cleaning, rinsing, disinfection, and vacuum drying into a single automated cycle.
  Interventions: Device: Pulsed Vacuum Cleaning and Disinfection Device
- Ultrasonic Cleaning Group (Active Comparator): A total of 400 rigid endoscopic instruments were cleaned using a conventional vacuum ultrasonic cleaner, followed by a separate spray cleaning and drying process, after manual pre-treatment.
  Interventions: Device: Vacuum Ultrasonic Cleaner

INTERVENTIONS:
Device: Pulsed Vacuum Cleaning and Disinfection Device — After manual pre-treatment, instruments were placed into the pulsed vacuum cleaning and disinfection machine (Shandong Xinhua Medical, Model PC-150L). The automated program included pulsed vacuum cleaning, rinsing, thermal disinfection (93°C for 2.5 minutes), and vacuum drying.
  Arms: Pulsed Vacuum Cleaning Group
Device: Vacuum Ultrasonic Cleaner — After manual pre-treatment, instruments were cleaned in a vacuum ultrasonic cleaner (Shandong Xinhua Medical, Model super-6000) with a multi-enzyme solution for a minimum of 5 minutes. This was followed by a separate process in a spray cleaning and disinfection machine for rinsing and drying.
  Arms: Ultrasonic Cleaning Group

SUMMARY:
This study is a prospective, comparative trial designed to evaluate the cleaning effectiveness of a novel pulsed vacuum cleaning and disinfection device against a conventional vacuum ultrasonic cleaner for rigid endoscopic instruments. Key outcomes measured include cleaning time, cleaning quality (via visual, light source, and ATP inspection), protein residue levels, and instrument damage rate.

DETAILED DESCRIPTION:
Rigid endoscopic instruments, due to their complex structure, pose significant challenges for cleaning and sterilization, which is critical for preventing hospital-acquired infections. Traditional methods like ultrasonic and spray cleaning have limitations in efficiency and thoroughness. This study was conducted to assess a newer technology, the pulsed vacuum cleaning and disinfection device, which integrates cleaning, rinsing, disinfection, and drying. A total of 800 rigid endoscopic instruments were divided into two groups: one cleaned with the pulsed vacuum device (Observation Group) and the other with a conventional vacuum ultrasonic cleaner (Control Group). The study aims to provide evidence-based insights into the efficiency, efficacy, and safety of the pulsed vacuum device for clinical application in sterilization supply centers.

ELIGIBILITY:
Inclusion Criteria:

* Rigid endoscopic instruments scheduled for post-operative cleaning.
* Types of instruments included: laparoscopes, hysteroscopes, arthroscopes, nephroscopes, prostate resection scopes, and thoracoscopes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Protein Residue Detection | Assessed once per instrument, immediately following the completion of the single cleaning procedure (Day 0)
  The level of residual protein on the instrument surface was measured using the biuret method. Outcomes were categorized as clean, mild, moderate, or severe contamination. The rate of clean instruments was compared between groups.
Cleaning Qualification Rate | Assessed once per instrument, immediately following the completion of the single cleaning procedure (Day 0)
  The cleaning effect was evaluated based on the "Hospital Sterilization Supply Center Part 3: Cleaning, Disinfection, and Sterilization Effect Monitoring Standards". Qualification was determined by a composite of three methods:
  * Visual Inspection: No visible contaminants.
  * Magnifying Light Source Observation: No visible stains or residues under magnification.
  * ATP Fluorescence Detection: Relative Light Unit (RLU) value ≤2000. The percentage of instruments passing all three checks was calculated.

SECONDARY OUTCOMES:
Cleaning Time | Assessed during a single time point event (the cleaning procedure on Day 0). The duration of the measurement is approximately 60 to 90 minutes.
  Total time required to process all 400 instruments in each group, from the start of manual pre-treatment to the completion of the final drying step. Unit: Minutes.
Instrument Damage Rate | Assessed at a single time point: immediately after the completion of the single cleaning procedure on Day 0.
  The number and percentage of instruments found to be damaged (e.g., deformation, breakage) after the complete cleaning and drying cycle in each group.

CONTACTS AND LOCATIONS:
Locations (1):
- Shijiazhuang Maternal and Child Health Hospital, Shijiazhuang, Hebei, China